CLINICAL TRIAL: NCT05801198
Title: Addressing Both Naturally Occurring and ACT-induced Plasmodium Reservoirs Using Artemisia Infusions to Accelerate Malaria Elimination and Eradication in Rwanda: A Proof of Concept Randomized Controlled Trial
Brief Title: Addressing Asymptomatic Plasmodium Reservoirs to Accelerate Malaria Elimination and Eradication in Rwanda.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: King Faisal Hospital Rwanda (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 452/RNEC/2022
Record Dates: First submitted 2023-03-01; First posted 2023-04-06 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-03

CONDITIONS: Malaria,Falciparum
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Artemisia Afra (Experimental): artemisia afra 10g/ day for 14 days
  Interventions: Dietary Supplement: Artemisia afra or Annua 10g oral infusion/tea per day for 14 days
- Artemisia Annua (Experimental): artemisia annua 10g/ day for 14 days
  Interventions: Dietary Supplement: Artemisia afra or Annua 10g oral infusion/tea per day for 14 days
- No treatment (No Intervention)

INTERVENTIONS:
Dietary Supplement: Artemisia afra or Annua 10g oral infusion/tea per day for 14 days — Participants will be recruited after completing standard malaria treatment, and those who have a positive qRT-PCR for plasmodium gametocyte reservoirs will be randomly assigned to either artemisia afra tea, or artemisia annua tea or into the control group with no intervention
  Arms: Artemisia Afra; Artemisia Annua

SUMMARY:
The investigators believe that to effectively achieve malaria elimination in Rwanda, it is critical to target the human reservoirs of Plasmodium falciparum using local and readily available Artemisia tea. Asymptomatic infections detectable by PCR are important reservoirs because they often persist for months and harbor gametocytes, the parasite stage infectious to mosquitoes. Lessons learnt from this study will be of critical importance for health decision makers with regard to potential malaria control. MSc and PhD students will be trained and the impact of this research project will be enormous on the socioeconomic transformation of Rwanda.

DETAILED DESCRIPTION:
According to the World Health Organization (WHO) world malaria 2021 report, there were 241 million cases of malaria in 2020, with 627 000 estimated deaths during the same year - an increase of 69 000 deaths over the previous year. The African continent continues to carry a disproportionately high share of the global malaria burden. In 2020 the Region was home to 95% of all malaria cases and 96% of deaths. Children under 5 years of age accounted for about 80% of all malaria deaths in the Region. Despite admirable progress in the first 15 years of this century, there has been setbacks with regard to achieving malaria elimination.

Malaria is a parasitic vector-transmitted infection caused by Plasmodium species. Four main human species are: P. falciparum, the most virulent and predominant specie in Sub-Saharan Africa, P. Ovale, P. vivax and P. malariae, and one zoonotic specie P. knowlesi. It is a disease responsible for catastrophic health and socio-economic impact mainly due to Plasmodium falciparum, which is responsible for substantial morbidity and mortality especially in children under five years and pregnant women.

When a Plasmodium-carrying Anopheles mosquito takes a blood meal on an individual, saliva is injected together with the sporozoites, which migrate to the liver, thereby beginning a cycle. Once humans become infected, the hepatic cycle lasts 10 to 14 days (in the case of P. falciparum), after which thousands of asexually reproducing merozoites are released into the peripheral blood where they invade and develop inside mature erythrocytes. The blood stage parasites are those that cause the symptoms of malaria. In a continuous pattern, during asexual replication in the blood stream, a small proportion of the parasites undergo sexual development that lasts approximately 10 days in the case of P. falciparum, resulting in the production of transmissible gametocyte forms. These gametocytes responsible for parasite transmission from humans to the mosquito vector, are insensitive to most conventional antimalarial drugs and are often long-lived (population lifespan of up to 55 days following successful antimalarial therapy), thereby ensuring malaria transmission over several weeks. Disrupting malaria transmission therefore requires the development of new anti-gametocyte drugs with safety profiles that allow for population-wide treatment campaigns.

Rwanda has made great strides during the last two decades by investing strategically in health system strengthening, increasing access to care by establishing community based health insurance, resulting in substantial declines in disease burden. However, since 2012, the country has been experiencing a persistent upsurge of malaria. From 2012 to 2018, malaria incidence increased significantly from 48 per 1000 to 403 per 1000, an almost 10x increase. By 2019-2020, the number of cases was reduced by more than half, to 198 per 1000. Although transmission is heterogeneous in Rwanda, the entire population is considered at risk of malaria. The primary Plasmodium (P.) species found in Rwanda, the agent responsible for this disease, is P. falciparum, but P. malariae and P. ovale have also been identified and this is mostly in the cosmopolitan main city of Kigali that receives frequent travelers and tourists.

Despite the gains made, recent upsurges and concerns about growing drug resistance calls for more dynamic, accessible, cost effective and adaptive mechanisms to combat, and potentially eliminate malaria all together. Over the past decade, several public health measures attempting to eradicate malaria were instituted, but this goal remains elusive to date and the country, and like most of sub-Saharan Africa, Rwanda continues to face a high burden of malaria mortality and morbidity.

In Rwanda, and many other African household setting, families frequently have both younger children and elderly grandparents living together. When a household member has Plasmodium reservoirs, this puts both the younger children and older more vulnerable family members at risk for recurrent severe malaria infections. The significance of asymptomatic household carriers in sustaining transmission of malaria was evidenced both in South East Asia and in Africa.

Malaria control measures that are currently deployed include the selective use of various WHO recommended strategies like control of mosquito breeding, timely diagnosis, and management of cases, as well as use of chemoprophylaxis for highly vulnerable population groups such as children under 5, pregnant women and visitors from non-endemic zones. This has provided some gains in reducing malaria burdens globally in recent years and, generating increased hopes for malaria elimination/eradication in the near future. However, such gains are severely threatened by the emergence and worldwide spread of both insecticide and antimalarial drug resistance. Resistance to Artemisinin combination therapy (ACTs), the first line treatment recommended by WHO is evident in Southeast Asia and has also been reported in African countries. Eliminating malaria will therefore necessitate the development of innovative approaches and tools, including new treatment options and vector control measures.

During 2021, the WHO recommended the use of the RTS, S/S2 malaria vaccine for the prevention of P. falciparum malaria in children living in regions with moderate to high transmission as defined by WHO. However, phase 3 trials showed relatively little efficacy, and the fact that the vaccine itself is unlikely to meet the goal of malaria eradication by itself. With further vaccine candidates in the pipeline that are being evaluated in vaccine trials, there is hope that alternative parasite targets and vaccination strategies will continue to be developed. Another recent positive is from combined RTS, S/S2 vaccine and chemoprevention that showed that this approach was non-inferior to chemoprevention alone in preventing uncomplicated malaria. The combination of these interventions resulted in a lower incidence of uncomplicated malaria, severe malaria, and death from malaria than each intervention alone.

More recently, a novel vaccine R21 has been undergoing phase 2 trials. Despite being similar to RTS, S2, it fuses together a hepatitis B antigen and half the circumsporozoite protein - a larger portion than in RTS, S2. The developers believed that this combination would be at least as effective as RTS, S, but less expensive. In a double-blind, randomized, controlled, phase 2b trial a low-dose circumsporozoite protein-based R21 vaccine, was given to children aged 5-17 months in Nanoro, Burkina Faso, with two different doses of adjuvant Matrix-M (MM). R21/MM appears safe and significantly immunogenic in this cohort of African children, and shows promising efficacy.

More vaccine trials have been conducted with radiation-attenuated Plasmodium falciparum sporozoite (PfSPZ) vaccine, hypothesized to provide protection against P. falciparum infection in malaria-naïve adults and children. Preclinical studies show that T cell-mediated immunity is required for protection and is readily induced in humans after vaccination. There was, however, no significant protection against P. falciparum infection in any dose group at 6 months which was the primary end point of the study.

Asymptomatic malaria is prevalent in endemic regions and throughout all seasons and identifying them often requires the use of highly sensitive diagnostic tools, including molecular approaches such as PCR. Eliminating malaria in areas with stable malaria transmission will therefore require the sustainable use of integrated vector-parasite approaches targeting both the human asymptomatic reservoirs and vector reservoirs, while paying attention to toxicity from drugs, and ensuring resistance is not further worsened.

Literature shows that asymptomatic reservoirs can be eliminated in mass treatment programs. In the past, diverse mass treatment strategies (Mass drug administration (MDA)) have been proposed and tried proving to rapidly reduce malaria particularly in regions with seasonal malaria transmission in parts of Africa and in China. Unfortunately, the use of ACTs in community-directed treatment of asymptomatic malaria poses a challenge, not only from drug resistance, but also the observation of potentiation of gametocyte proliferation upon ACT administrations. Contrarily to the above reported challenges of ACTs to be used in MDA, in vitro studies demonstrated that Artemisia annua and Artemisia afra infusions or powdered leaves were efficacious, where both clearly demonstrated potent inhibition of parasitemia and gametocytemia. It has also been shown that Artemisia annua contains not only artemisinin but also other components that demonstrate a synergistic complex anti-malaria effect. Artemisia afra does not contain any artemisinin. In a recent human double-blind clinical trial and in other previous studies both plants were reported to stably cure malaria, including ACT-resistant cases as well as killing transmissible gametocyte forms. Their chemo protective potential was also observed in these and other studies.

We believe that to effectively achieve malaria elimination in Rwanda, it is critical to target the human reservoir of P. falciparum using local and readily available Artemisia infusions. Asymptomatic infections detectable by PCR are an important reservoir because they often persist for months and harbor gametocytes, the parasite stage infectious to mosquitoes.

III. Research objectives General objective; To provide a proof of concept that Artemisia infusions, both annua and afra, are efficient and sufficient to eliminate residual Plasmodium reservoirs following malaria treatment. The investigators will determine the current prevalence of human Plasmodium reservoirs in our community and in our post malaria treated patients, both the wild type, and mutated/resistant strains at King Faisal Hospital and associated health facilities. We will further determine those associated with mutation in the Kelch13 gene or other candidate genes implicated in treatment failure.

Specific objectives;

1. Provide a proof of concept that Artemisia infusions are efficient and sufficient to empty human Plasmodium reservoirs in asymptomatic volunteers in community and following malaria treatment.
2. Investigate P. falciparum household clusters in Under Five old malaria patients as well as in individuals infected with strains carrying mutations associated with resistance to treatment, and explore how engineering a Malaria Family Registry can be used as a tool for better disease control in Rwanda
3. To assess the safety of Artemisia afra and Artemisia annua by monitoring urine chemistry tests, kidney (urea, creatinine and electrolytes), and liver function tests (transaminases, bilirubin).
4. To investigate the prophylactic potentials of Artemisia infusions once reservoirs have been cleared.
5. Assess utilization and acceptability of Artemisia herbal medicine in Rwandan communities.
6. Study the socio-economic impact of human Plasmodium reservoir drainage in Rwandan community.

IV. Methodology

Study setting The study will be conducted on patients seeking medical care for malaria at King Faisal Hospital, associated health facilities, CHUB, as well as in the community targeting asymptomatic Plasmodium carriers.

Study design The study will be conducted as a proof of concept open randomized controlled trial using permuted block randomization/random varying sizes. The investigators will recruit at least 125 participants within 14 days following completion of standard malaria treatment. Patients will be asked to sign informed consent and a PCR/RT-PCR will be performed to test for P. falciparum reservoirs. We will use a Real Time PCR (qPCR) cut off cycle threshold (CT value) above or equal to 40, which has been established based on negative African control and European controls that have never been exposed to malaria before. Blood samples from the recruited participants will also be investigated for single nucleotide polymorphisms (SNPs) in the Kelch13 gene by sequencing the propeller domain of this gene within which point mutations associated with Artemisinin resistance have been reported. In case of absence of SNP in K13, the search for other gene mutation associated with treatment failure will be done by whole genome sequencing and further addressed by laboratory parasite culture assays. From the screened participants, one hundred (100) with residual parasites (induced reservoirs) will then be assigned into 3 groups: two intervention groups and 1 control group

Sample size determination The investigators are planning a study of independent cases and controls with 1 control for 2 cases. Preliminary data indicates that the failure rate among controls is ≥ 0.75. If the true failure rate for treated subjects is ≤ 0.25, we need to study at least 40 treatment subjects and 20 controls in order to detect such a difference with a 95% power at a 0.05 significance level. We will thus require 40 patients in each intervention group and 20 controls, a total of 100. For us to randomize 100, we plan to screen at least 125 patients during our set recruitment period. Based on the fact that under 5 children are the most vulnerable with the highest malaria associated mortality and morbidity and will not participate in our clinical trials, we will recruit them as index cases for our household clusters survey. Household members of these children will thus be screened using PCR to establish status of plasmodium reservoirs and to ascertain if there are any mutations of significance within the plasmodium circulating in the home. Confirmed reservoirs in adult household members who consent will be treated with Artemisia tea.

Study population For the clinical approach, the study will recruit adults between 18 and 65 years for the Artemisia tea proof of concept intervention between 15th April 2023 until 30th June 2026. However, based on the fact that under 5 children are the most vulnerable with the highest mortality, the under 5 post malaria treated children will be included as index cases for our household clusters survey and family registry development. Although children will not be included during this initial proof of concept study, we intend to develop galenic formulations appropriate to pediatric age group at a later stage.

For de community approach, asymptomatic household members will be screened using PCR/RT-PCR to establish status of Plasmodium reservoirs and to ascertain if there are any mutations within the residual Plasmodium circulating in the home. Based on this, a family registry around the young children index cases will be built as a tracking tool, and Artemisia tea given to the adults with a goal to eliminate the household cluster reservoirs. We will then track over at least a 6 months' period to see if any differences in children whose household clusters were treated with the infusions and those who were not with regard to malaria infections. This will be tested as an additional potential malaria surveillance and control measure.

To further investigate if Artemisia infusions could possess prophylactic potential, we intend to pursue the study with the already enrolled participants by changing the posology. The 75% of participants with reservoir emptied will be randomized in 3 groups: the first group of 12 participants will proceed with Artemisia tea one cup (335 ml) of 10g/L (A. afra) or 10g/L (A. annua) every day; the second group of 12 participants will receive Artemisia tea one cup (335 ml) of 10g/L (A. afra) or 10g/L (A. annua) once every week; the last group of 6 participants will be the controls. If the Artemisia infusions with either A. afra or A. annua block Plasmodium reservoir fill up in more than 75% of the participants compared to less than 25% of controls, then the study will have a 95% power to detect a difference between the prophylactic group and the controls at a significance level of 0.025.

To monitor for toxicity, kidney and liver function tests will be investigated at the beginning and after 14 days of Artemisia tea, as well as monthly during the prophylactic phase of at least 6 months.

To address acceptability and impact of the research interventions, appropriate surveys will be conducted.

Data management and analysis All data will be handled using standard confidentiality principles and managed with EpiInfo and analyzed using STATA 17 software packages. Participants will be described based on their socio-demographic characteristics as means and standard deviations for continuous variables or proportions for categorical variables. An intention-to-treat (ITT) analysis using two sample proportion will be used to determine the chances of the plasmodium reservoir being emptied. Survival analysis with cox regression will be carried out to evaluate the plasmodium reservoir emptying time and time for recrudescence / reinfection. Data will be compared between groups using either the Chi-square or Fischer exact test after checking for the smallest expected value. Mean change from baseline Means will be compared using either a parametric (student t or ANOVA) or a non-parametric (Mann-Whitney/Wilcoxon or Kruskal-Wallis) test after checking for normality of distribution and equality of variances.

Ethical considerations All study participants will have a detailed explanation about the study and requested to freely sign a written informed consent. Ethics clearance has been approved by the Rwanda National Ethics committee (120/RNEC/2022 May 2022, Amended October 2022). Rwanda Food and Drug Authority clearance application has been initiated.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed as asymptomatic reservoir of Plasmodium in the community or after completing standard malaria treatment.
* Leave for at least one month in Rwanda for non-national
* Be between 18 and 65 years of age, and in good general health.
* Not taking any other malaria drug for prevention or treatment.
* Children 5 years and above will be recruited as index cases for household cluster survey.

Exclusion Criteria:

* Have known hypersensitivity to any ingredients of the test treatment.
* Have participated in any other malaria drug trial or device less than 14 days before.
* History or presence of clinically significant medical, psychiatric, or emotional condition that would compromise the safety of the subject or adherence to the interventional requirements.
* Be pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Negative RT-PCR for plasmodium reservoirs | 14 days
  The primary outcome will be negative P. falciparum blood stage infection as detected by RT-qPCR (CT ≥ 40) after 14 days of Artemisia infusion treatment.

SECONDARY OUTCOMES:
urea and creatinine | 14 days
  Kidney function test will be done on serum, to establish a baseline, and repeated at day 14 following completion of the treatment
Liver enzymes; ALT/ AST | 14 days
  Baseline test of the liver transaminases will be done on serum, and repeated at day 14
Urine dipstick | 14 days
  a urine dipstick will be done; PH, leucocytes, blood, nitrites, specific gravity, ketones, glucose, urobilinogen.

IPD SHARING:
Plan to Share IPD: Yes
By publication in relevant scientific journals
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 36 months
Access Criteria: Authorization will be provided by study sponsors